CLINICAL TRIAL: NCT01166334
Title: WebQuit Online Smoking Cessation Study
Acronym: WebQuit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Jonathan Bricker, PhD, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FHCRC IR#7181
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Smoking
Keywords: Smoking; Smoke; Cigarette; Cessation; Quit; Online; Web; Stop
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- WebQuit study group (Active Comparator): Intervention arm 1 (identity and description withheld to protect integrity of study)
  Interventions: Behavioral: WebQuit study group
- WebQuit control group (Active Comparator): Intervention arm 2 (identity and description withheld to protect integrity of study)
  Interventions: Behavioral: WebQuit control group

INTERVENTIONS:
Behavioral: WebQuit study group — Description withheld to protect integrity of study
  Arms: WebQuit study group
Behavioral: WebQuit control group — Identity and description withheld to protect integrity of study
  Arms: WebQuit control group

SUMMARY:
Would you like to quit smoking?

Seattle's Fred Hutchinson Cancer Research Center is launching a new study that may be able to help. Participants who enroll in this study will be randomly assigned by computer (like flipping a coin) to one of two online programs. The goal of this study is to learn which of these programs is the most effective at helping people stop smoking. Findings from this study will be used to help build more effective online smoking cessation programs in the future.

Participants in both of the smoking cessation programs used in this study will receive:

* Interactive tools for dealing more effectively with urges to smoke
* Step-by-step guides for quitting smoking
* Personalized plans for quitting and remaining smoke-free
* Electronic links for reaching one-on-one expert help for quitting

Participants will be asked to complete online questionnaires, including a brief three-month follow-up survey.

There is no cost for participating in this study.

To enroll in this study or for more information, please visit www.webquit.com.

This study is being conducted by Seattle's Fred Hutchinson Cancer Research Center (www.fhcrc.org), a world leader in advancing the prevention, diagnosis and treatment of cancer. The principal investigator for the WebQuit smoking cessation study is Dr. Jonathan Bricker, a faculty member at both the Hutchinson Center and at the University of Washington in Seattle.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* a current resident of the US
* someone who has smoked daily for at least the past 12 months
* someone who wants to quit smoking in the next 30 days
* willing and able to read in English
* able to connect to the Internet for at least one hour per week for three consecutive months
* able to use a website
* not participating in other smoking cessation interventions
* willing and able to complete a Baseline Survey
* willing to be randomized to either online program

Exclusion Criteria:

* inability to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence | 3 months and 6 months post treatment
  No smoking in the past 7 days, as reported 3 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Kwon DM, Santiago-Torres M, Mull KE, Sullivan BM, Bricker JB. Older adults who smoke: Do they engage with and benefit from web-based smoking cessation interventions? Prev Med. 2022 Aug;161:107118. doi: 10.1016/j.ypmed.2022.107118. Epub 2022 Jun 17. PMID 35718119
- [Derived] Jones HA, Heffner JL, Mercer L, Wyszynski CM, Vilardaga R, Bricker JB. Web-based acceptance and commitment therapy smoking cessation treatment for smokers with depressive symptoms. J Dual Diagn. 2015;11(1):56-62. doi: 10.1080/15504263.2014.992588. PMID 25671683